CLINICAL TRIAL: NCT07028086
Title: Prospective, Multicenter, Single-Arm Clinical Study of Mitoxantrone Liposome Combined With Azacitidine and Venetoclax in the Treatment of Secondary AML, AML With Extramedullary Involvement, and Myeloid Sarcoma
Brief Title: VAM in Secondary AML, AML With Extramedullary Involvement, and Myeloid Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Shen yang, Chief physician, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAVEN_01
Record Dates: First submitted 2025-06-04; First posted 2025-06-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia; Myeloid Sarcoma
Keywords: Secondary AML; AML with Extramedullary Involvement; Myeloid Sarcoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Sarcoma, Myeloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MAVEN_GROUP (Experimental)
  Interventions: Drug: VAM_GROUP

INTERVENTIONS:
Drug: VAM_GROUP — Mitoxantrone Liposome 24mg/m², IV, administered as a single dose or divided doses at the investigator's discretion based on the patient's condition; Azacitidine 75mg/m², IV drip, Day 1 to Day 7; Venetoclax 100mg on Day 1, 200mg on Day 2, and 400mg on Day 3 to Day 14.

SUMMARY:
The mitoxantrone liposomal enhances the tissue permeability of mitoxantrone by incorporating liposomal groups compared to the conventional mitoxantrone formulation, while also reducing the concentration of free mitoxantrone, thereby minimizing drug side effects-particularly cardiotoxicity.

Building upon this, the investigators aim to investigate the efficacy and safety of the liposomal mitoxantrone hydrochloride injection in patients with secondary AML, AML with extramedullary involvement, or myeloid sarcoma, in order to explore alternative therapeutic strategies for these populations.

ELIGIBILITY:
Inclusion Criteria:

1. The patient fully understands this study, voluntarily participates, and signs the informed consent form (ICF)
2. Age 18-65 years
3. Clinically diagnosed, previously untreated acute myeloid leukemia (non-APL), meeting any one of the following criteria: a. Secondary acute myeloid leukemia; b. Therapy-related acute myeloid leukemia; c. AML with extramedullary/myeloid sarcoma; d. Age ≥60 years, assessed as fit-AML;
4. Normal cardiac function, with left ventricular ejection fraction (LVEF) ≥50%
5. Liver and kidney function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal (ULN) (≤5 times ULN for patients with liver involvement); total bilirubin ≤1.5 times ULN; serum creatinine ≤1.5 times ULN
6. Eastern Cooperative Oncology Group (ECOG) performance status score: 0-2

Exclusion Criteria:

1. Assessed as unfit- or frail-AML;
2. Patients with a history or concurrent diagnosis of other malignancies requiring treatment
3. Uncontrolled systemic diseases (e.g., advanced active infections, uncontrolled hypertension, etc.)
4. Known history of immediate or delayed hypersensitivity reactions to the same class of study drugs or excipients
5. Pregnant or breastfeeding women, or patients who refuse to use effective contraception during the study period
6. Patients with a history of severe neurological or psychiatric disorders
7. Other severe medical conditions, such as myocardial infarction, severe or unstable angina, severe arrhythmias
8. Cerebrovascular events (including transient ischemic attacks), etc.
9. Known infection with human immunodeficiency virus (HIV); active hepatitis B or C infection; inactive hepatitis carriers or subjects with low viral titers after receiving non-prohibited antiviral therapy are not excluded
10. Subjects who have received strong or moderate CYP3A inducers/inhibitors or strong P-gp inhibitors or related foods within 7 days before starting the study treatment
11. Patients unable to take oral medications or with malabsorption syndrome
12. Patients deemed by the investigator to be unsuitable for participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Composite Complete Remission Rate | After completing two cycles (each cycle is 28 days) of VAM therapy

SECONDARY OUTCOMES:
Event-Free Survival | from data of AML diagnosis until the data of events, assessed up to 2 years
Overall Survival | from enrollment to study completion, a maximum of 2 years
Safety: Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | During the two cycles (each cycle is 28 days) of VAM therapy and follow-up for 2 years after completion

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes